CLINICAL TRIAL: NCT07374016
Title: Evaluation of a Training Recommendation Strategy for Trail Runners.
Acronym: TRAILWISE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 24CH251
Record Dates: First submitted 2026-01-21; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Endurance Training
Keywords: Trail running; Performance; Training recommendations; Artificial intelligence

STUDY DESIGN:
Intervention Model Description: Longitudinal, controlled, randomised, prospective study by downloading training data and questionnaires via smartphone.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GEN: generic training plan group (Active Comparator): The GEN group will follow a generic training plan that will be created from a platform that is both free and popular, offering training plans for trail-running (The Decathlon Pacer application).
  Interventions: Procedure: Training recommendations GEN
- PERSO: non-adaptive personalized group (Active Comparator): The PERSO group will follow a plan that takes into consideration the training history, in particular the number of hours per week over the previous two years; the runner's level; age and sex; time available for training; and access to mountainous terrain.
  Interventions: Procedure: Training recommendations PERSO
- PERSO-ADAPT group: adaptive personalized group (Experimental): The PERSO-ADAPT group will include the same information as the PERSO group, but the training will also be adapted on a weekly basis according to the following feedback: state of fatigue assessed by questionnaire and heart rate variability; state of overtraining, assessed by questionnaire; degree of session completion).
  Interventions: Procedure: Training recommendations PERSO-ADAPT

INTERVENTIONS:
Procedure: Training recommendations GEN — Generic training plan that will be created from a platform that is both free and popular, offering training plans for trail-running (The Decathlon Pacer application).
  Arms: GEN: generic training plan group
Procedure: Training recommendations PERSO — A training plan that takes into account the rider's training history, in particular the number of hours per week over the last two years, the rider's level, age and gender, the time available for training and access to mountainous terrain.
  Arms: PERSO: non-adaptive personalized group
Procedure: Training recommendations PERSO-ADAPT — A training plan that takes into account the rider's training history, in particular the number of hours per week over the last two years, the level, age and gender of the rider, the time available for training and access to mountainous terrain. Training will also be adapted on a weekly basis according to the following feedback: state of fatigue assessed by questionnaire and heart rate variability; state of overtraining, assessed by questionnaire; degree of completion of sessions.
  Arms: PERSO-ADAPT group: adaptive personalized group

SUMMARY:
Finding the optimal training, i.e. the training that enables the athlete to achieve the best performance while preserving their physical and psychological integrity, is a multi-factorial issue.

Each individual's background and training capacity are very different, hence the need for personalised training. The availability of data combined with advances in Artificial Intelligence (data modelling and analysis sciences, big data, machine learning, deep learning, etc.) offer the opportunity to refine our understanding of training and adapt recommendations according to the runner's profile for a given objective (achieving a time over a distance, completing an event, etc.). The strategy that the investigators wish to evaluate as part of this trial could make it possible to recommend an optimal training load, as well as the distribution of intensities (as a percentage of the aerobic threshold, anaerobic threshold, VVO2max, etc). The two features are (i) the personalisation will be based on training history, the level of the runner, age and gender, and the runner can focus on training, and (ii) the strategy will be adaptive, i.e. the algorithm will update the training load in real time based on contextual data about the athlete (level of fatigue via heart rate variability, feedback on recent training sessions, feelings of stress).

ELIGIBILITY:
Inclusion Criteria:

* Have no contraindications to trail running (Fédération Française d'Athlétisme test procedures)
* Have been trail running competitively for at least 1 year
* In possession of an ITRA performance index
* Intends to run at least one ITRA-indexed race in the second half of the follow-up period
* Own a training watch, and intend to record all training sessions of more than 10 minutes in their shared database
* Have freely given their written consent.

Exclusion Criteria:

* Any person with chronic joint pathologies (e.g. recurrent sprains, patellar or ligament problems) or cardiac pathologies.
* Any person with chronic or central neurological pathologies.
* Any person deprived of their liberty or under legal protection (guardianship, curatorship, safeguard of justice, family habilitation).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1209 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of the ITRA performance index | Month : 10
  The main criterion for assessing the improvement in trail running performance will be the increase in the ITRA performance index of users following PERSO-ADAPT compared with the increase in the ITRA score of PERSO and GEN. The ITRA Performance Index (PI) is a tool that estimates a runner's level of performance. The performance index can be used to compare the level of different trail runners around the world and is built on a scale up to a maximum of 1000 points. The top of the scale corresponds to the theoretical best possible level.

SECONDARY OUTCOMES:
Number of injuries | Weeks : 1 to 40
  The number of injuries will be assessed on the basis of weekly injury records, with injury defined as any physical pain or disability resulting from running that prevents running for at least one day.
ROF (Rating-of-Fatigue Scale) | Weeks : 1 to 40
  Fatigue will be assessed each week using the ROF (Rating-of-Fatigue Scale), validated in French. This scale from 0 to 10 with a pictogram gives an assessment that best reflects the perception of fatigue at that precise moment (from 0: not at all tired to 10: completely tired and exhausted).
RPE (Rating of Perceived Exertion) | Weeks : 1 to 40
  RPE (Rating of Perceived Exertion) will be assessed each week using the Borg scale and a visual analogue scale (VAS). It comprises 11 levels of perceived exertion, ranging from 0 (no exertion) to 10 (maximum exertion).
Hooper questionnaire | Weeks : 1 to 40.
  Overtraining will also be assessed using the Hooper questionnaire. The higher the score, the more likely the athlete is to be in a state of physical or mental overload.
The '36-12' field test | Weeks : 6, 13, 20, 27, 34, 40.
  Objective performance will be assessed by measuring critical speed, obtained using the '36-12' field test. This test, which can take the place of a training session, is carried out on a training track which is usual for the runner, and consists of: a run of 3600 metres, 30 minutes recovery time, then a run of 1200 metres. The time will be measured for each of the runs and the heart rate continuously recorded using the classic training heart rate monitor.
The 1200 test | Weeks : 6, 13, 20, 27, 34, 40.
  Objective performance will be assessed through changes in the duration of the 1200 test: after a 10-minute low-intensity warm-up, the participant will have to run 1200 m on a track at an intensity considered to be "low", recording his speed and heart rate at the same time using his watch.

CONTACTS AND LOCATIONS:
Overall Officials: Leonard FEASSON, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Unités de Myologie et de Médecine du Sport, Saint-Etienne, France, France

IPD SHARING:
Plan to Share IPD: No